CLINICAL TRIAL: NCT05775653
Title: Group-based [ADAPT] Versus One-to-one [Usual] Occupational Therapy for Improving Activities of Daily Living in People With Chronic Conditions: A Protocol for a Randomized Controlled Pilot and Feasibility Study (The Go:OT Trial)
Brief Title: Group-based [ADAPT] Versus One-to-one [Usual] Occupational Therapy: A Pilot and Feasibility Study
Acronym: Go:OT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parker Research Institute (Other)
Collaborators: Rehabilitation Center Rødovre Municipality (Genoptræning Rødovre Kommune) (Unknown); Den Kommunale Kvalitetsudviklingspulje (Unknown); Lundbeckpuljen (Unknown); Oak Foundation (Other); Tværspuljen (Unknown)
Responsible Party: Principal Investigator, Eva Ejlersen Wæhrens, Professor, Parker Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Parker Institute
Record Dates: First submitted 2023-02-23; First posted 2023-03-20 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2023-11

CONDITIONS: Chronic Condition; Chronic Conditions, Multiple
MeSH Terms: conditions — Chronic Disease; Multiple Chronic Conditions

STUDY DESIGN:
Intervention Model Description: A randomized controlled pilot and feasibility study
Who Masked: Participant, Outcomes Assessor
Masking Description: The trial attempts to blind clients and assessors. Clients are informed that they will be allocated to one of two occupational therapy intervention programs that both aims to improve ADL ability, but overall primarily differ in the format i.e. a group-based versus a one-to-one intervention program. Clients are however not informed, which of the two types of formats that are the new experimental intervention format (ADAPT). Baseline assessments are conducted prior to randomization by the local project coordinator and the project coordinator is instructed not to reveal which intervention that is the new experimental intervention. The post- and follow-up assessor, an externally recruited occupationa therapist from a nearby hospital research unit, is also instructed not to disclose which intervention that is the new. Finally, all clients are reminded not to disclose any details, that may provide the outcome assessor with insight regarding their group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADAPT program (Experimental): The ADAPT program is a structured and individualized group-based program.
  Interventions: Other: ADAPT program
- Usual Occupational Therapy (UOT) (Active Comparator): UOT is delivered by one occupational therapist. .
  Interventions: Other: UOT

INTERVENTIONS:
Other: ADAPT program — The ADAPT program is a structured and individualized group-based program, in which two occupational therapists teach groups of people the skills of problem-solving more efficiently as means to overcome ADL task performance problems. The ADAPT program 3.0 includes 10 two-hour sessions and is followed by two booster sessions to support sustainable gains.
  Arms: ADAPT program
Other: UOT — UOT is delivered by one occupational therapist. Sessions are individualised and focus on improving ADL ability e.g. by practicing the performance of ADL task. UOT typiccally includes 7 one-to-one sessions of 60 minutes, delivered over a 10-week period in the clients´ homes. The dose is however not fixed but based on the occupational therapists´ clinical judgement.
  Arms: Usual Occupational Therapy (UOT)

SUMMARY:
Background: The number of people living with chronic conditions limiting the ability to perform activities of daily living (ADL) tasks is increasing. Occupational therapists are trained to deliver interventions to improve ADL ability. Municipality occupational therapy interventions are usually delivered as one-to-one sessions in the client´s home. While this intervention format might be effective, a group-based intervention format might be as effective but more cost-effective? Hence, the group-based ADAPT program was developed, piloted and evaluated for its functioning and feasibility in municipality settings. These studies provided initial evidence for the ADAPT Programs effectiveness. A randomized controlled trial (RCT) is however needed to document effectiveness, processes, and cost-effectiveness of the ADAPT program versus usual occupational therapy (UOT) for people with chronic conditions. Prior to the RCT, this pilot and feasibility study will be conducted to test aspects of trial design, conduct and processes as well as intervention content and delivery.

Material and Methods: A total of 16 home dwelling persons with chronic conditions, experiencing ADL task performance problems will be randomized and allocated to receive ADAPT (intervention) or UOT (control). Effectiveness and cost-effectiveness assessments are collected at baseline and post intervention i.e., 3-months (week 12) and 6-months (week 26) from baseline. Pilot and feasibility aspects will be evaluated by means of registrations forms filled out by the OTs delivering ADAPT and people with chronic conditions attending ADAPT. Registrations are designed to inform aspects of 1) recruitment and retention, 2) trial participation, 3) impact of trial on participants and staff, 4) completion rates, 5) fidelity and dose 6) assesable information and 7) adaptation of trial conduct to local context. Progression criteria for when to 'go', 'amend' or 'be alert/stop' are defined, to support the decision on whether to continue to RCT or the need to adjust design or procedures,

DETAILED DESCRIPTION:
TThe specific aims of this pilot and feasibility study are to evaluate:

1. how recruitment procedures work and if participants accept randomization (recruitment and retention)
2. if clients feel adequately informed about the purpose of the assessments done and the content and time use regarding interventions delivered (trial participation)
3. if trial participation has unanticipated impacts on ADAPT OTs (e.g. workload) (Impact of trial on staff)
4. if registration forms and outcome measurements are completed (Completion rates)
5. the extent of which the ADAPT OT adhere to the ADAPT program manual and deliver key components within each session (fidelity and dose)
6. if data informing about intervention delivered in UOT is accessible from client records (Assessable information)
7. if ADAPT OTs perceive organizational factors to facilitate or hinder program delivery (adaptation of trial conduct to local context)?

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* ≥ one year since medical diagnosed with one or more chronic conditions
* Lives in own home
* Experience ADL task performance problems
* Show ADL motor ability measures <1.50 on the AMPS ADL motor skills scale (indicate increased effort during ADL task performance)
* Communicate independently and relevantly orally and in writing (without severe cognitive deficits, aphasia, significant hearing loss or dyslexia)
* Willing and interested in attending occupational therapy interventions focused on improving ADL task performance.

Exclusion Criteria:

* ADL process ability measures <0.00 indicating that the person is unlikely to profit from educational programs focused on using adaptational strategies
* Mental illness and/or other acute (<3 months) conditions effecting ADL task performance
* Language barriers
* Known substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-11-09 (Actual)

PRIMARY OUTCOMES:
Change in observed motor ability | week 12
  Assessment of Motor and Process Skills (AMPS) is a unidimensional linear measure in which higher scores are better outcome

SECONDARY OUTCOMES:
Change in self-reported ability to perform activities of daily living tasks | week 12 and 26
  ADL-Interview (ADL-I, Performance) is a unidimensional linear measure in which higher scores are better outcome
Change in observed motor ability | week 26
  Assessment of Motor and Process Skills (AMPS) is a unidimensional linear measure in which higher scores are better outcome
Change in observed process ability | week 12 and 26
  Assessment of Motor and Process Skills (AMPS) is a unidimensional linear measure in which higher scores are better outcome
Change in self-reported satisfaction with ability to perform activities of daily living tasks- | week 12 and 26
  ADL-Interview (ADL-I Satisfaction)
Perceived change in ability to perform activities of daily living tasks | week 12 and 26
  Transition Questionnaire (TRANS-Q) based on a scale of seven categorical variables
Perceived change in occupational balance | week 12 and 26
  Transition Questionnaire (TRANS-Q) based on a scale of seven categorical variables
Perceived change ability to problemsolve | week 12 and 26
  Transition Questionnaire (TRANS-Q) based on a scale of seven categorical variables
Perceived change in need for assistance | week 12 and 26
  Transition Questionnaire (TRANS-Q) based on a scale of seven categorical variables
Perceived change in Quality fo life | week 12 and 26
  Transition Questionnaire (TRANS-Q) based on a scale of seven categorical variables
Perceived Quality of life | week 12 and 26
  EuroQoL 5 dimensions (EQ-5D) based on a scale of five categorical variables
Perceived generel health | week 12 and 26
  First questions in the MOS 36-item Short Form Survey Instrument based on a scale with 5 categorical variables

OTHER OUTCOMES:
Perceived mental well-being | week 12 and 24
  WHO-5 questionnaire based on a 6-point ordinal scale in which higher is better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Cecilie von Bülow, PhD, Principal Investigator — Parker Institute, Bispebjerg and Frederiksberg Hospital
Locations (1):
- The Parker Research Institute, Department of Rheumatology, Copenhagen University Hospital, Bispebjerg and Frederiksberg Frederiksberg, Denmark, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: No